CLINICAL TRIAL: NCT05403762
Title: Comparison of Two Skin Protection Regimes for the Prevention of Incontinence-associated Dermatitis in Geriatric Care: an Exploratory Trial (PID)
Brief Title: Prevention of Incontinence-associated Dermatitis
Acronym: PID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Prof. Dr. Jan Kottner, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PID; 01KG2020 (Other Grant/Funding Number: German Federal Ministry of Education and Research (BMBF))
Record Dates: First submitted 2022-05-23; First posted 2022-06-03 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Incontinence-associated Dermatitis
Keywords: Skin care; Long-term care; Nursing home resident; Erythema; Geriatric medicine
MeSH Terms: conditions — Erythema

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ESENTA™ Skin Barrier Spray (Experimental): In the intervention group I, standardized mild skin cleansing regimen and daily topical application of a film-forming skin protectant at the exposed skin areas will be applied by nursing staff.
  Interventions: Other: ESENTA™ Skin Barrier Spray (ConvaTec, UK)
- Hydrophobes Basisgel DAC (Experimental): In the intervention group II, standardized mild skin cleansing regimen and daily topical application of a hydrophobic skin protectant at the exposed skin areas will be applied by nursing staff.
  Interventions: Other: Hydrophobes Basisgel DAC
- Standard Care (No Intervention): In the control group, standardized mild skin cleansing regimen without application of an additional skin protectant will be conducted by nursing staff.

INTERVENTIONS:
Other: ESENTA™ Skin Barrier Spray (ConvaTec, UK) — The skin protectant will be applied on clean and dry skin exposed to urine and stool. After application, the solvent evaporates leaving a silicone film on the skin surface.
  Other Names: Film-forming skin protectant
  Arms: ESENTA™ Skin Barrier Spray
Other: Hydrophobes Basisgel DAC — The skin protectant will be applied on clean and dry skin. It contains 95% paraffin oil and creates a hydrophobic layer on the skin surface.
  Other Names: Hydrophobic skin protectant
  Arms: Hydrophobes Basisgel DAC

SUMMARY:
Incontinence-associated dermatitis (IAD) is an inflammation of the skin caused by prolonged direct contact of the skin with urine and/or stool. Elderly and care-dependent people are often affected by this type of inflammation. Gentle skin cleansing and the use of skin protection products are recommended. Available skin protection products can be categorized into film-forming or lipophilic skin protectants depending on the ingredients and overall composition. There is no evidence about the superiority of one product compared to another regarding skin protection. The overall aim of this study is to compare the effects of two skin protection products compared to an untreated control group. An exploratory trial in elderly nursing home residents and geriatric patients will be conducted.

DETAILED DESCRIPTION:
Incontinence-associated dermatitis (IAD) is an inflammation of the skin caused by prolonged and direct contact of the skin with urine and/or stool. It may occur in all age groups but elderly and care-dependent incontinent people are often affected by this type of inflammation. Promotion of continence, use of absorbent products and structured skin care are recommended to prevent and/or treat IAD. Available skin protection products can be categorized into film-forming or lipophilic skin protectants depending on the ingredients and overall composition. Currently, there is no evidence about the superiority of one product compared to another regarding skin protection. The overall aim of this study is to compare the effects of two skin protection products compared to an untreated control group. An exploratory randomized controlled trial in incontinent elderly nursing home residents and geriatric patients will be conducted. In the two intervention groups, a film-forming or a lipophilic skin protection product will be applied in addition to standardized skin care regimens. Every other day, investigators will perform skin inspections, including instrumental skin measurements to quantify erythema for a total study period of n= 14 days. IAD- related pain and itch will be assessed. A total of n= 210 nursing home residents and geriatric patients in Berlin, Germany, aged over 65 years, who are affected by urinary and faecal incontinence without signs of severe IAD will be included.

ELIGIBILITY:
Inclusion Criteria:

* Geriatric patients or residents being incontinent of urine and stool
* Expected minimum length of stay of 14 days at the care facility
* Intact skin with no clinical signs of IAD OR
* intact skin with early clinical signs of IAD (IAD category 1A)
* Written informed consent

Exclusion Criteria:

* Residents/patients at the end of life
* Residents/Patients with IAD category 1B, 2A, 2B and/or signs of clinical infection in the IAD area
* Any skin condition or wounds (at investigational areas of the skin) requiring additional treatment (e. g. pressure ulcers, intertrigo, infection)
* Known hypersensitivity or allergy to silicones and/or topical leave-on products
* Topical treatments in the IAD area.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2022-08-19 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of incontinence-associated dermatitis (IAD) | 14 Days
  Number of subjects developing IAD of all subjects (cumulative incidence).
  Classification of IAD according to Ghent Global IAD Categorisation Tool (GLOBIAD) (Category 1A, 1B, 2A, 2B). The GLOBIAD categorises IAD severity based on visual inspection of the affected skin areas.
  Category 1A: Persistent redness without clinical signs of infection Category 1B: Persistent redness with clinical signs of infection Category 2A: Skin loss without clinical signs of infection Category 2B: Skin loss with clinical signs of infection
Erythema (instrumental measurement) | 14 Days
  Erythema measured with the Mexameter MX® 18 (Courage + Khazaka, Cologne, Germany). Means of two duplicate measurements per skin area are displayed in arbitrary units (AU) ranging from 0 (= no erythema) to 999 (= extreme erythema).
Erythema (visual inspection) | 14 Days
  Clinical rating of erythema is conducted according to the item 'Redness' of the incontinence-associated dermatitis and its severity (IADS) instrument. The 3-Item-Scale describes 'Redness' as (1) none, (2) pink, (3) red/ bright red.
Incidence of erosion | 14 Days
  The presence (no or yes) of erosion is defined according to the latest International League of Dermatological Societies glossary of cutaneous lesions as a loss of either a portion of or the entire epidermis. Number of subjects developing erosions of all subjects (cumulative incidence).
Incidence of maceration | 14 Days
  The presence (no or yes) of maceration is defined as the result of prolonged exposure (of the skin) to moisture and causes the skin to soften and breakdown so that the connective fibres can be teased apart and the skin often exhibits a white appearance. Number of subjects developing maceration of all subjects (cumulative incidence).
IAD related pain | 14 Days
  To assess pain, a Numeric Rating Scale (NRS) is applied. That scale ranges from 0 (= no pain) to 10 (= worst possible pain) for patients/residents without cognitive impairment (according to Mini-Mental-State-Examination (MMSE) with scores of 24 or higher).
Patient satisfaction | 14 Days
  To assess patient satisfaction, a Numeric Rating Scale (NRS) is applied.That scale ranges from 0 (= dissatisfied) to 10 (= very satisfied) for patients/residents without cognitive impairment (according to Mini-Mental-State-Examination (MMSE) with scores of 24 or higher).
Incidence of IAD related itch | 14 Days
  IAD related itch will be reported directly by patients (yes or no). Number of subjects reporting itch of all subjects (cumulative incidence).
Presence of local intolerances | 14 Days
  The presence of local intolerances will be assessed with the following options:
  (0) None;
  1. homogeneous redness with scattered papules;
  2. homogeneous redness and homogeneous infiltration
  3. homogeneous redness and infiltration with vesicles
  4. homogeneous redness and infiltration with coalescing vesicles
Adverse Events (AEs) and Serious Adverse Events (SAEs) | 14 Days
  AEs and SAEs will be documented and reported according to the current regulation (EU) 2017/745 of the European Parliament and of the Council of 5 April 2017 on medical devices (MDR) Article 2.
Incidents and serious incidents | 14 Days
  Incidents abd serious incidents will be documented according to the definition of the EU regulation 2017/745 MDR Article 2 and reported to the Bundesinstitut für Arzneimittel und Medizinprodukte (BfArM).

CONTACTS AND LOCATIONS:
Overall Officials: Jan Kottner, Prof., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol will be shared as part of this trial registration.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Anonymized IPD will be made available beginning 12 months and ending 36 months after publication of trial results.
Access Criteria: IPD will be shared with researchers who submit a methodologically sound proposal. The proposal must clearly state the research objectives and the intended methods of analysis. It is planned to share the data with restricted access via zenodo.org.

REFERENCES:
- [Derived] El Genedy-Kalyoncu M, Fastner A, Volzer B, Raeder K, Neumann K, Lahmann NA, Kottner J. Comparison of two skin protection regimes for the Prevention of Incontinence-associated Dermatitis in geriatric care (PID): a study protocol for an exploratory randomised controlled pragmatic trial. BMJ Open. 2022 Sep 29;12(9):e065909. doi: 10.1136/bmjopen-2022-065909. PMID 36175092